CLINICAL TRIAL: NCT05679869
Title: Effects of Natural Sounds on Attention Restoration in Virtual Reality
Acronym: VEARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Ministry of National Development, Singapore (Other Government); Housing and Development Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Georgios CHRISTOPOULOS, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COT-V4-2020-1-S005
Record Dates: First submitted 2022-09-05; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Fatigue; Mental Fatigue; Behavioral Performance; Heart Rate Variability; Working Memory
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Simulated Outdoor Environment (Active Comparator): Exposure to recorded outdoor environmental sounds
  Interventions: Other: No masking sound
- VR Simulated Outdoor Environment with Masking Sounds (Experimental): Exposure to recorded outdoor environmental sounds augmented with masking sounds
  Interventions: Other: Masking Sound

INTERVENTIONS:
Other: Masking Sound — Prerecorded environmental noise and masking sounds played from headphones
  Arms: VR Simulated Outdoor Environment with Masking Sounds
Other: No masking sound — Prerecorded environmental noise but no masking sounds played from headphones
  Arms: VR Simulated Outdoor Environment

SUMMARY:
This study aims to examine whether listening to natural sounds in a noisy virtual reality environment compared to no natural sounds influences physiological markers.

DETAILED DESCRIPTION:
The investigators hypothesize that listening to natural sounds has restorative effects on attention by supporting greater use of involuntary attention. This generates the prediction that exposure to natural sounds in the context of a noisy environment will have greater restorative effects on attention (i.e., physiological) as compared to the control group (exposed to noise only). Individual differences (i.e., age, gender, caffeine and food intake, body mass index, skin temperature, noise sensitivity, sleep quality, baseline physiology and behavioural performance) will be examined and accounted for.

ELIGIBILITY:
Inclusion Criteria:

* Singapore-based
* Non-clinical
* 18-35years

Exclusion Criteria:

* Individuals with hearing difficulties or failing to meet the minimal threshold for normal hearing
* Individuals with a history of ear, developmental, neurological, or psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | 1 day (during fatiguing task and sound intervention)
  Electrocardiograph (Change)
Change in Fatigue State Questionnaire | baseline, up to 2 mins after fatiguing task and up to 2 mins after sound intervention
  Change in Fatigue State Questionnaire Score

CONTACTS AND LOCATIONS:
Locations (1):
- Cultural Science Innovations, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No